CLINICAL TRIAL: NCT05467150
Title: Maternal Probiotic Supplementation for Improved Neurodevelopmental Outcomes in Infants of Diabetic Mothers (IDMs)
Brief Title: Maternal Probiotic Supplementation for Improved Outcomes in Infants of Diabetic Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2022-29947
Record Dates: First submitted 2022-06-16; First posted 2022-07-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infant of Diabetic Mother
Keywords: infant of diabetic mother; probiotic; gut microbiome; neurodevelopment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Supplement (Experimental): Participants (mothers) randomized to this arm will take one Culturelle® Digestive Daily Probiotic Capsule per day from study enrollment through the first postpartum month. Each capsule contains 10 billion CFU of Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: Probiotic Supplement
- No intervention (No Intervention): Participants (mothers) randomized to this arm will agree to continue not taking any over the counter probiotic supplements from study enrollment through the first postpartum month.

INTERVENTIONS:
Dietary Supplement: Probiotic Supplement — The probiotic that will be used is Culturelle® Digestive Daily Probiotic Capsules. Each capsule contains 10 billion CFU of Lactobacillus rhamnosus GG (LGG).
  Arms: Probiotic Supplement

SUMMARY:
The purpose of this study is to test the hypothesis that maternal probiotic supplementation is associated with infant gut microbiome variation and improved neurodevelopmental outcomes as measured by ERP performance in infants of diabetic mothers (IDMs), a cohort that is at-risk for recognition memory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people in their second or third trimester with a diagnosis of gestational diabetes.
* BMI 18.5-45 kg/m2 at first prenatal visit
* Age 21-45 at time of delivery
* Report social support for and intention to exclusively breastfeed for at least 3 months
* Singleton pregnancy

Exclusion Criteria:

* Alcohol consumption >1 drink per week during pregnancy/lactation
* Tobacco consumption during pregnancy/lactation
* Inability to speak/understand English
* Known congenital metabolic, endocrine disease (other than GDM), or congenital illness affecting infant feeding
* History of type I Diabetes
* Birthing parent currently taking over the counter probiotic preparation

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Infant auditory recognition ERP performance at 1 month: P200 amplitude | 1 month of age
  At one month of age, an auditory recognition memory ERP will be performed. Components of interest will be the P200 amplitude (in microvolts) The P200 is a positive component of the ERP waveform and a measure of early perceptual processing of stimuli.
Infant auditory recognition ERP performance at 1 month: Negative slow wave difference score | 1 month of age
  At one month of age, an auditory recognition memory ERP will be performed. Components of interest will be latency in milliseconds. The area under the curve of the negative slow wave (NSW, a late slow-resolving component if the ERP waveform, which is thought to index detection of a novel stimulus against the background of familiar stimuli).
Infant visual recognition ERP performance at 6 months: Slow wave difference score | 6 months of age
  At 6 months of age, visual-evoked potential ERP paradigms will be performed. We will be measuring the latency and amplitude of the N290, a negative component occurring between 150-400ms (representing face processing), the amplitude of the negative central (NC) component, occurring between 350-700ms and thought to index attention, and the area under the curve of the slow-resolving positive component occurring between 900-1500ms that indexes memory updating.
Infant VEP performance at 6 months: latency to peak of P100 | 6 months of age
  The main component of interest in the VEP waveform is a large positive wave peaking at about 100 ms (P100). We will be looking at the latency to the peak of the P100 component (milliseconds) as a measure of speed of processing.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States